CLINICAL TRIAL: NCT02273518
Title: A Double-blind, Randomised, 3-way Cross-over Study to Compare the Pharmacokinetics of Dipyridamole in Three Different Asasantin ER Extended Release (ER) 200 mg Dipyridamole/25 mg ASA Formulations in Healthy Male and Female Volunteers
Brief Title: Study to Compare the Pharmacokinetics of Dipyridamole in Three Different Asasantin Extended Release (ER) Formulations in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 9.144
Record Dates: First submitted 2014-10-23; First posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (3):
- Asasantin ER, new formulation I (Experimental)
  Interventions: Drug: Asasantin ER, new formulation I
- Asasantin ER, new formulation II (Experimental)
  Interventions: Drug: Asasantin ER, new formulation II
- Asasantin ER, present commercial formulation (Active Comparator)
  Interventions: Drug: Asasantin ER, present commercial formulation

INTERVENTIONS:
Drug: Asasantin ER, new formulation I
  Arms: Asasantin ER, new formulation I
Drug: Asasantin ER, new formulation II
  Arms: Asasantin ER, new formulation II
Drug: Asasantin ER, present commercial formulation
  Arms: Asasantin ER, present commercial formulation

SUMMARY:
Comparative pharmacokinetics of dipyridamole in two new formulations of Asasantin ER compared to the present commercial formulation

ELIGIBILITY:
Inclusion Criteria:

* All participants in the study should be healthy males or females, range from 21 to 50 years of age and be within ± 20 % of their normal weight (Broca-Index)
* Prior to admission to the study all volunteers will have given, in accordance with good clinical practice (GCP) and the local legislation, their written informed consent
* Subsequently each subject will have his medical history taken and will receive a complete medical examination (incl. blood pressure and pulse rate measurements) as well as a 12-lead ECG
* Hematopoietic, hepatic and renal function tests will be carried out in the laboratory
* The subjects will fast for 12 hours before collection of specimens for all laboratory evaluations
* The above mentioned examinations will be performed within 14 days before the first administration of the test substance

Exclusion Criteria:

* Volunteers are excluded from the study if the results of the medical examination or laboratory tests are judged by the clinical investigator to differ significantly from normal clinical values
* Subjects with known gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Subjects with diseases of the central nervous system (such as epilepsy) or with psychiatric or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Subjects with chronic or relevant acute infections
* Subjects with allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Volunteers who have taken a drug with a long half-life (≥ 24 hours) within one month or less than ten half-lives of the respective drug before enrolment in the study
* Volunteers who receive any other drugs which might influence the results of the trial during the week previous to enrolment in the study
* Volunteers who participate in another study with an investigational drug within the last two months preceding the study
* Volunteers who are unable to refrain from smoking on study days
* Volunteers who smoke more than10 cigarettes (or equivalent) per day
* Volunteers who drink more than 60 g of alcohol per day
* Volunteers who are dependent on drugs
* Volunteers who donate blood (≥ 100 mL) within the last four weeks
* Volunteers who participate in excessive physical activities within the last week before the study (e.g. competitive sports)
* Volunteers who suffer from any other disease or abnormality of clinical relevance
* History of hemorrhagic diatheses
* History of gastro-intestinal ulcer, perforation or bleeding
* History of bronchial asthma
* History of glucose-6-phosphate dehydrogenase (G-6-PD) deficiency

Female subjects:

* Pregnancy
* Positive pregnancy test
* No adequate contraception (adequate contraception e.g. sterilization, intrauterine devices (IUD), oral contraceptives)
* Inability to maintain this adequate contraception during the whole study period
* Lactation period

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2001-04; Primary Completion 2001-05 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of dipyridamole in plasma at steady state (AUC,ss) | Up to 48 hours after start of drug administration
Percent peak trough fluctuation of dipyridamole in plasma (%PTF) | Up to 48 hours after start of drug administration

SECONDARY OUTCOMES:
Maximum concentration of the analytes in plasma at steady state (Cmax,ss) | Up to 48 hours after start of drug administration
Minimum measured concentration of the analytes in plasma at steady state over a uniform dosing interval τ (Cmin,ss) | Up to 48 hours after start of drug administration
Time from dosing to the maximum measured concentration of the analytes in plasma at steady state over a uniform dosing interval τ Time from dosing to the maximum measured concentration of the analytes in plasma at steady state (tmax,ss) | Up to 48 hours after start of drug administration
Percent area under the curve fluctuation of the analytes in plasma (AUCfluct) | Up to 48 hours after start of drug administration
Terminal half-life of the analytes in plasma (t1/2) | Up to 48 hours after start of drug administration
Percent of dose of the analytes recovered unchanged in urine (Ae%) | Up to 24 hours after start of drug administration
Ratio of peak concentration of the analytes in plasma over area under the curve at steady state (Cmax,ss / AUC,ss) | Up to 48 hours after start of drug administration
Number of subjects with clinically relevant changes in vital signs (blood pressure, pulse rate) | up to 8 days after last study drug administration
Number of subjects with clinically relevant changes in 12-lead ECG | up to 8 days after last study drug administration
Number of subjects with clinically relevant changes in laboratory values | up to 8 days after last study drug administration
Number of subjects with adverse events | up to 8 days after last study drug administration